CLINICAL TRIAL: NCT02751294
Title: A Randomized, Open-label, Single-period, Parallel-group Study in Healthy Subjects to Determine the Effects of Dissolution Profile on the Pharmacokinetics (Via Both Venous and Peripheral Micro-samples) of Single Oral 300 mg Doses of Tafenoquine (SB-252263) Tablets + 30 mg Tafenoquine Stable Isotope Labelled (SIL) Solution
Brief Title: A Study to Assess the Effects of Dissolution Profile on the Pharmacokinetics of Single Oral Doses of Tafenoquine Tablets and Tafenoquine Stable Isotope Labelled Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Medicines for Malaria Venture (Other); Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201780
Record Dates: First submitted 2016-04-21; First posted 2016-04-26 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Malaria, Vivax
Keywords: Healthy Volunteer; Malaria; Pharmacokinetics; Tafenoquine
MeSH Terms: conditions — Malaria, Vivax; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TQ Control+ TQ SIL (Experimental): Subjects received TQ Control product (2 tablets) and 30 mg TQ SIL solution orally with water after a meal.
  Interventions: Drug: Tafenoquine Control; Drug: Tafenoquine SIL
- TQ X + TQ SIL (Experimental): Subjects received 2 tablets of Tafenoquine dissolution profile X and 30 mg TQ SIL solution orally with water after a meal.
  Interventions: Drug: Tafenoquine dissolution profile X; Drug: Tafenoquine SIL

INTERVENTIONS:
Drug: Tafenoquine Control — It will be supplied as a dark pink, capsule-shaped, film-coated tablet plain on both sides containing 150 mg tafenoquine
  Arms: TQ Control+ TQ SIL
Drug: Tafenoquine dissolution profile X — It will be supplied as a dark pink, capsule-shaped, film-coated tablet plain on both sides containing 150 mg tafenoquine and will be "intermediate aged TQ Product".
  Arms: TQ X + TQ SIL
Drug: Tafenoquine SIL — It will be compounded at site and will be administered as 0.3 mg/mL (100mL to be dosed, equivalent to 30 mg) aqueous Solution of SIL Tafenoquine.

SUMMARY:
This study will investigate the effect of Tafenoquine (TQ) 150 mg tablet ageing (dissolution profiles) on human exposure of TQ comparing the relative bioavailability of TQ from tablets exhibiting different dissolution profiles in healthy subjects. This is a single-centre, 2-arm, randomized open-label, parallel-group study in healthy subjects. All subjects will arrive in the unit approximately 24 hours prior to dosing and will be discharged after the 72-hour post-dose assessments are completed. Subjects will return for outpatient visits on Days 7, 14, 21, 28, and 56 after dosing. A total of 14 subjects (n=7 subjects in each arm) are planned to be enrolled. All subjects will receive a single dose of study medication (2x150 mg TQ tablets + 30 mg TQ SIL in solution) and participate through a 56-day post dose follow-up visit. To enable the application of peripheral microsampling in planned paediatric studies, a comparison of the measured pharmacokinetic (PK) exposure via peripheral blood collection (via microsampling) to venous collection will also be performed in this study.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Between 18 and 55 years of age inclusive, at the time of signing the informed consent
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator and the GlaxoSmithKline (GSK) Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Subject values outside the normal range should always be excluded from enrolment.
* Body weight between >=35 kilogram (kg) and <=100 kg.
* Male subjects only.
* Capable of giving signed informed consent as described in study protocol, which includes compliance with the requirements and restrictions listed in the consent form and in the study protocol

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Alanine Aminotransferase (ALT) and bilirubin >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) > 450 millisecond (msec) Note: The QTc is the QTcF). Other calculation methods (e.g. QT interval corrected using Bazett's formula [QTcB], QTcF) machine-read or manually over-read are not acceptable.
* Use of prescription (except acetaminophen at doses of 2 grams/day) or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 30 days of the study defined as: an average weekly intake of >14 drinks for males. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 millilitre [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Positive results for drugs of abuse as mentioned in protocol.
* Cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 30 days prior to screening.
* History of sensitivity to TQ, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* History of thalassaemia; or current or past history of methemoglobinemia or methemoglobin percentage above the reference range at screening.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* The subject has been dosed with TQ within 10 months prior to being dosed in this study.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 15 days of dosing with TQ or matched-placebo.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Subjects with a hemoglobin values outside the lower limit of normal range. A single repeat is allowed for eligibility determination.
* Documented phenotypic Glucose-6-phosphate dehydrogenase (G6PD) deficiency, determined by a quantitative assay of enzyme activity. Defined as <70% of locally defined median.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Ratio of the geometric means for the area under plasma concentration-time curve (AUC) for Tafenoquine X | Samples will be collected at Pre-dose and 1, 2, 6, 9, 12, 15, 20, 24, 36, 48, 60, and 72 hours post dose on Day 1 and single sample on Day 7, 14, 21, 28, and 56
  Blood samples for PK analysis of TQ will be collected for evaluation of ratio of the geometric means (90% Confidence Interval [CI]) for the area under plasma concentration-time curve from 0 to time t (AUC [0-t]) and area under the concentration-time curve from 0 to infinity (AUC[0-inf]) for the treatment group dissolution profile X compared to Control.

SECONDARY OUTCOMES:
Safety as assessed by clinical monitoring of blood pressure | Up to 12 hours
  Systolic and diastolic blood pressure will be measured in semi-supine position after approximately 5 minutes rest. Blood pressure will be measured at pre-dose (at least 30 min. prior to dosing and at least 15 min. after waking) and at 12 hours post dose.
Safety as assessed by clinical monitoring of pulse rate | Up to 12 hours
  Pulse rate will be measured in semi-supine position after approximately 5 minutes rest. Pulse rate will be measured at pre-dose (at least 30 min. prior to dosing and at least 15 min. after waking) and at 12 hours post dose.
Safety as assessed by clinical monitoring of electrocardiogram (ECGs) | Day -1
  Single 12-lead ECGs will be obtained in the semi-supine position at screening using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT interval corrected for heart rate according to Fridericia's formula (QTcF) intervals
Safety as assessed by clinical monitoring of Haematology parameters | Up to Day 14
  Haematology parameters include Platelet Count, red blood cell (RBC) Indices, white blood cell (WBC) count with differential, RBC Count, mean cell volume (MCV), neutrophils, hemoglobin, mean corpuscular hemoglobin (MCH), lymphocytes, hematocrit, monocytes, methemoglobin %, eosinophils and basophils. It will be assessed on Day -1, Pre-dose and post-dose at Day 7 and Day 14.
Safety as assessed by clinical monitoring of Clinical Chemistry parameters | Up to Day 14
  Clinical chemistry parameters includes blood urea nitrogen, potassium, aspartate aminotransferase (SGOT), total and direct bilirubin, creatinine, sodium, alanine aminotransferase (SGPT), total protein, glucose, calcium, alkaline phosphatase and albumin. It will be assessed on Day -1, Pre-dose and post-dose at Day 7 and Day 14.
Safety as assessed by clinical monitoring of Urinalysis parameters | Up to Day 14
  Urinalysis parameters include specific gravity, pH, glucose, protein, blood and ketones. It will be assessed on Day -1, Pre-dose and post-dose at Day 7 and Day 14
Number of participants with adverse events (AE) | Up to Day 63
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal.
Area under the plasma concentration-time curve from time 0 to last measurable concentration (AUC0-t) for Tafenoquine | Samples will be collected at Pre-dose and 1, 2, 6, 9, 12, 15, 20, 24, 36, 48, 60, and 72 hours post dose on Day 1 and single sample on Day 7, 14, 21, 28, and 56
  PK samples will be obtained from venous blood and peripheral blood collection (via microsampling)
Maximum plasma concentration (Cmax) for Tafenoquine | Samples will be collected at Pre-dose and 1, 2, 6, 9, 12, 15, 20, 24, 36, 48, 60, and 72 hours post dose on Day 1 and single sample on Day 7, 14, 21, 28, and 56
  PK samples will be obtained from venous blood and peripheral blood collection (via microsampling)
Time to Cmax (tmax) for Tafenoquine | Samples will be collected at Pre-dose and 1, 2, 6, 9, 12, 15, 20, 24, 36, 48, 60, and 72 hours post dose on Day 1 and single sample on Day 7, 14, 21, 28, and 56
  PK samples will be obtained from venous blood and peripheral blood collection (via microsampling)
Terminal half-life (t1/2) for Tafenoquine | Samples will be collected at Pre-dose and 1, 2, 6, 9, 12, 15, 20, 24, 36, 48, 60, and 72 hours post dose on Day 1 and single sample on Day 7, 14, 21, 28, and 56
  PK samples will be obtained from venous blood and peripheral blood collection (via microsampling)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Goyal N, Mohamed K, Rolfe K, Sahota S, Ernest T, Duparc S, Taylor M, Casillas L, Koh GCKW. Application of the Stable Isotope Label Approach in Clinical Development-Supporting Dissolution Specifications for a Commercial Tablet Product with Tafenoquine, a Long Half-life Compound. AAPS J. 2018 Jun 4;20(4):74. doi: 10.1208/s12248-018-0234-5. PMID 29869298